CLINICAL TRIAL: NCT06198491
Title: Evaluation of Educational Interventions Targeting Beliefs About Human Papillomavirus (HPV) Among Female Employees
Brief Title: Evaluation of Educational Interventions Targeting Beliefs About Human Papillomavirus (HPV)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Selva Dilan Golbasi Koc, Director, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E-80558721-050.99-413737
Record Dates: First submitted 2023-12-25; First posted 2024-01-10 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Beliefs; HPV; Education, Medical; Intervention
Keywords: Belief; HPV; Education; Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training for HPV misbeliefs 1 (Experimental): Participants will receive misbeliefs about HPV; training where misbeliefs are mentioned before the current information.
  Interventions: Behavioral: Misbeliefs about HPV training
- Training for HPV misbeliefs 2 (Experimental): Participants will receive misbeliefs about HPV; training where misbeliefs are mentioned after the current information.
  Interventions: Behavioral: Misbeliefs about HPV training

INTERVENTIONS:
Behavioral: Misbeliefs about HPV training — Intervention trainings mentioned false beliefs before or after the current knowledge

SUMMARY:
The goal of this clinical trial is to compare the effects of two different educational training programs on beliefs about Human Papillomavirus (HPV) in a group of female hospital employees. The main questions it aims to answer are: • Within the scope of the study, are the training programs provided to reduce misconceptions about HPV effective? • Which educational program is more effective in reducing misconceptions about HPV? Participants will • Complete a pre-test online the day before the first training date to determine the level of their misconceptions about HPV. • Receive informative messages via Whatsapp once a day for three days according to the training program they are assigned to. • Repeat the pre-test at the end of the training programs and one month later. • Receive the more effective training program after one month after the test repetition for the control group. Researchers will compare "Misbeliefs about HPV" and "Current Knowledge about HPV" titled training programs on reducing misconceptions about HPV.

DETAILED DESCRIPTION:
The human papillomavirus (HPV) can cause health problems ranging from warts in the mouth or genital area to cervical, vaginal, vulvar, penile and anal cancers. Some beliefs about diseases or infectious agents have a negative impact on the early diagnosis and treatment of diseases, particularly by increasing the stigmatization effect of sexually transmitted diseases. Features such as the fact that mucosal contact is sufficient for transmission, that infected people can be symptom-free for a long time, that cancer often develops slowly, and that there are similarities with other sexually transmitted viruses such as HIV (human immunodeficiency virus) or herpes can have a negative impact on knowledge and beliefs about HPV.

It is known that it is crucial to emphasize correct information, not to repeat or point out inaccuracies when taking action to combat false beliefs or myths. In the context of the COVID-19 pandemic, the importance of this approach has been frequently emphasized in the guidance contained in the confirmatory information on misinformation and disinformation. In our study, we want to compare the effectiveness of education models in which false beliefs or myths about HPV are conveyed before or after the current information.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Age >18 years and older
* Those who agree to participate in the study

Exclusion Criteria:

* Age <18 years
* Those who not agree to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Health Beliefs about Human Papillomavirus (HPV) | From enrollment to the end of intervention at 4 weeks
  Measuring with: "False Beliefs About HPV Scale"

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University Public Health Department, Odunpazari, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in beliefs about Human Papillomavirus. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As of March 2024
Access Criteria: "Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact selvadilangolbasi@gmail.com"